CLINICAL TRIAL: NCT03643523
Title: Prospective Study on the Determination of Albumina as an Early Predictor of Anastomotic Leak and Postoperative Infectious Complications in Colorectal Surgery
Brief Title: Determination of Albumina as an Early Predictor of Postoperative Infections in Colorectal Surgery
Acronym: ALB-CIR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Mora-Lopez, Doctor, Corporacion Parc Tauli
Other Study IDs: ALB-CIR
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Albumin; Double
Keywords: anastomitic leak, infectious complications, colorectal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALbumin level: Detection of serum albumin levels in postoperatory of colorectal surgery
  Interventions: Diagnostic Test: Albumine detection

INTERVENTIONS:
Diagnostic Test: Albumine detection — Control of serum albumine levels in postoperatori of colorectal surgery

SUMMARY:
Colorectal surgery has traditionally been associated with significant morbidity and prolonged hospital stay. Overall complication rates have been reported to be 26-35%. Infectious complications, in particular, represent a major cause of morbidity and mortality after colorectal surgery. Postoperative intra-abdominal infections after colorectal surgery are mainly due to anastomotic leakage. They occur in 5 to 15% of patients and carry a short term mortality of around 20%. They also have a major impact on the outcome of surgery as they prolong in hospital stay, increase treatment costs and worsen long-term survival in cancer patients. If diagnosed early, they can be treated effectively and their impact on surgery outcome is thus minimised.

There is a growing interest to find a biological marker useful for early detection of anastomotic leak; such a marker could play a pivotal role in the modern fast-track multimodal protocols, allowing safe and early discharge of patients after colorectal surgery.

Although C reactive protein (CRP) and procalcitonin (PCT) have been proposed as predictors for adverse outcomes in colorectal surgery, they both display the critical limitations of slow kinetics. Conversely, serum albumin (ALB) is a maintenance protein that is rapidly down regulated by inflammatory signals. There some studies about the use of postoperative ALB drop as a marker of predictor for clinical outcome. These studies are either retrospective or mix patients with different types of surgical procedures performed.

This study aimed to test the hypotheses that early postoperative albumin drop can predict anastomotic leaks and also can predict postoperative infectious complications earlier than other biological markers.

DETAILED DESCRIPTION:
Colorectal surgery (CS) has traditionally been associated with significant morbidity and prolonged hospital stay 1,2. Overall complication rates have been reported to be 26-35%.3,4,5,6 Infectious complications represent a major cause of morbidity and mortality after CS.6 Postoperative intra-abdominal infections after CS are mainly due to anastomotic leak (AL).7,8 They occur in 5 to 15% of patients and carry a short term mortality of around 20%.3 They also have a major impact on the outcome of surgery as they prolong in-hospital stay, increase treatment costs and worsen long-term survival in cancer patients.9,10,11 If diagnosed early, they can be treated effectively and their impact on surgery outcome is thus minimised.9 It is well-known that clinical features are not accurate predictors of AL in gastrointestinal surgery. 12,13 The white blood cell count is an unreliable predictor of either intra-abdominal infection or global postoperative infections. Routine imagine for the detection of leaks is not cost-effective and carries the drawback of radiation. Is it therefore essential to identify an early marker of infection, particularly in the era of "fast track" or "enhanced recovery " surgery, in which patients are discharged from hospital soon after operation, with the risk of intra-abdominal infection becoming evident after discharge thus inducing readmissions and late management.14 Althouhg early diagnosis of AL is a key point in reducing its clinical consequences in terms of morbidity and mortality, currently, AL diagnosis is often late because of misdiagnosis of medical complications and false-negative radiological examinations.15,16 Although C reactive protein (CRP) and procalcitonin (PCT) have been proposed as predictors for adverse outcomes in CS, they both display the critical limitations of slow kinetics.17,18,19 Conversely, serum albumin (ALB) is a maintenance protein that is rapidly down regulated by inflammatory signals. , Preliminary data suggested that ALB level rapidly dropped after surgery and correlated to outcomes in oesophageal, oral cancer, abdominal20 pancreatic, liver resection /trasplant and cardiac surgeries. However, prospective validation is missing, and ALB is not used to assess surgical stress or to predict outcomes.

Protein metabolism is significantly disturbed after any kind of traumatic event, for example, surgery, sepsis, and burn injuries , ALB has been identifyed as a reliable indicator of this process.21 Plasma concentration of ALB reveal an important decrease as early as a few hours after the hit.21,22,23 A previous studies estimated that 77% of the postoperative ALB decrease was due to redistribution, while 18% and 6% were attributed to blood loss and catabolism, respectively.24 Of note, transcapillary exchange rate early depended on the underlying trauma and no increase was noted after minor surgery.25,26 After operation, proinflamatory cytokines increase because of surgical stress, which leads to the reaction of circulating acute phase proteins, such as CRP and inteleukin-6, which have been widely use to predict complications after colorectal surgery.20 ALB, which is a marker of nutritional status and a negative acute phase protein, decreases immediately after surgery because of the physiological response to trauma. Increased capillary leakage of ALB is also one of the features of the systemic inflammatory response to surgical stress, which leads to a decreased level of plasma albumin. The response of ALB to surgical stress might occur earlier than CRP because ALB has quick kinetics after surgery.

There some studies about the use of postoperative ALB drop as a marker of predictor for clinical outcome. The first one, Hübner and col.21 shows a prospective pilot study about 70 patients undergoing frequent abdominal procedures of different magnitude. They measured ALB, CRP and CPT once daily starting the day before surgery until postoperative day (POD) 5. The conclusion of the estudy was that early postoperative ALB drop appeared to reflect the magnitud of surgical trauma and was correlated with adverse clinical outcomes. The group continues the same line of work and publishes another prospective cohort study with 138 patients undergoing major abdominal surgery. They collect blood samples before and on POD 0,1,2 and 3. They compare ALB decrease and CPR and CPT. The postoperative outcomes of the study were complications and length of hospital stay. They found a decrease of ALB of 10% yielded a sensitivity of 77.1% and a specificity of 67.2% (AUC : 78.3%) to predict complications. On the other hand, they also found that decrease of ALB of 10% on POD1 showed a threefold increased risk of overall postoperative complications.21 Antoher group, Ge et al.27 made a retrospective study about 626 patients undergoing major colorectal surgery with the main outcome were to identify risk factors for postoperative complications and to identify the factors associated with the ALB decrease. This study revealed the patients with a greater relative decrease in serum ALB in POD 2 were at higher risk of postoperative complications, prolonged postoperative hospital stays, an more Surgical Site infeccions after colorectal surgery. A cutoff value of 15% reduction in serum ALB on POD 2 distinguished patients at low risk and high risk for postoperative complications in an earlier stage and was more accurate the CRP level on POD 3 and 4.

These are the preliminary data that lead us to start our study in order to demonstrate the utility of the postoperative decrease of serum albumin as an early detector of anastomotic leak and infectious complications in patients undergoing major colorectal surgery This study aimed to test the hypotheses that early postoperative albumin drop can predict anastomotic leaks and also can predict postoperative infectious complications earlier than other biological markers

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients undergoing major colorectal surgery (expected to last 2 hours or more)
* Performing primary anastomosis
* Scheluded surgery
* Patients who give their written informed consent

Exclusion Criteria:

* Patients not meeting inclusion criteria at any time during the study (surgeries lasting less than 2 hours or anastomosis not performed. urgent surgery, not give written informed consent) will be excluded.

No other inclusion or exclusion criteria have been considered, however, the investigator should consider any circumstance where the benefit-risk for the patient is not adequate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on scheludec colorectal surgery with primary anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of serum albumine levels | One year

IPD SHARING:
Plan to Share IPD: No